CLINICAL TRIAL: NCT05106855
Title: Comparative Study of Immediate Single Unit Helix GM - Neodent Implants in Early Loading Protocols, With or Without Acqua Surface and With or Without Low Level Laser Photobiomodulation (LLLT). Single-blind Randomized Clinical Trial.
Brief Title: Comparative Study of Immediate Single Unit Implants in Early Loading Protocols, With or Without Photobiomodulation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Santiago de Compostela (Other)
Responsible Party: Principal Investigator, Mario Pérez Sayáns, Professor, University of Santiago de Compostela
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RCT-NEO-PBM-21
Record Dates: First submitted 2021-10-15; First posted 2021-11-04 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Dental Implant; Tooth Absence; Tooth Extraction
Keywords: immediate implant; post-extraction implant; early loading; photobiomodulation; oral rehabilitation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Implants GM Acqua surface, with LLLT. (Other): Surgical protocol Periotomes will be used for atraumatic extraction and/or a stainless steel tooth extractor.
  The implant, GM Acqua, will be placed in a flapless manner through the alveolus, manually or mechanically, and a minimum length of 2 mm longer than the root length. The implant placement site will be prepared following the manufacturer's protocol.
  The minimum torque that to be employed to attain primary stability of the implant will have to be ≥ 30 Ncm measured with a manual torque wrench. (Neodent®).
  After the implant has been placed, a healing abutment GM (Neodent®) will be placed, with a maximum torque of 10 N.cm.
  LLLT protocol:
  With a infrared diode laser, wavelength of 808 nm, continuous mode, a dose of 2J per spot, for 20 seconds per spot, the following irradiation protocol shall be applied: immediately after surgery and on days 3 and 7 after surgery, 4 spots (2 in the vestibular and 2 in lingual/palatal of the alveolus/implant).
  Interventions: Radiation: Low Laser Radiation; Procedure: Implant placement immediately after tooth extraction; Procedure: Installing the dental crown with early loading
- Implants GM Acqua surface, without LLLT. (Other): Surgical protocol Periotomes will be used for atraumatic extraction and/or a stainless steel tooth extractor.
  The implant, GM Acqua, will be placed in a flapless manner through the alveolus, manually or mechanically, and a minimum length of 2 mm longer than the root length. The implant placement site will be prepared following the manufacturer's protocol.
  The minimum torque that to be employed to attain primary stability of the implant will have to be ≥ 30 Ncm measured with a manual torque wrench. (Neodent®).
  After the implant has been placed, a healing abutment GM (Neodent®) will be placed, with a maximum torque of 10 N.cm.
  Interventions: Radiation: Low Laser Radiation off; Procedure: Implant placement immediately after tooth extraction; Procedure: Installing the dental crown with early loading
- Implants GM NeoPoros surface, with LLLT. (Other): Surgical protocol Periotomes will be used for atraumatic extraction and/or a stainless steel tooth extractor.
  The implant, GM NeoPoros, will be placed in a flapless manner through the alveolus, manually or mechanically, and a minimum length of 2 mm longer than the root length. The implant placement site will be prepared following the manufacturer's protocol.
  The minimum torque that to be employed to attain primary stability of the implant will have to be ≥ 30 Ncm measured with a manual torque wrench. (Neodent®).
  After the implant has been placed, a healing abutment GM (Neodent®) will be placed, with a maximum torque of 10 N.cm.
  LLLT protocol:
  With a infrared diode laser, wavelength of 808 nm, continuous mode, a dose of 2J per spot, for 20 seconds per spot, the following irradiation protocol shall be applied: immediately after surgery and on days 3 and 7 after surgery, 4 spots (2 in the vestibular and 2 in lingual/palatal of the alveolus/implant).
  Interventions: Radiation: Low Laser Radiation; Other: Changing the implant surface; Procedure: Implant placement immediately after tooth extraction; Procedure: Installing the dental crown with early loading
- Implants NeoPoros surface, without LLLT. (Other): Surgical protocol Periotomes will be used for atraumatic extraction and/or a stainless steel tooth extractor.
  The implant, GM NeoPoros, will be placed in a flapless manner through the alveolus, manually or mechanically, and a minimum length of 2 mm longer than the root length. The implant placement site will be prepared following the manufacturer's protocol.
  The minimum torque that to be employed to attain primary stability of the implant will have to be ≥ 30 Ncm measured with a manual torque wrench. (Neodent®).
  After the implant has been placed, a healing abutment GM (Neodent®) will be placed, with a maximum torque of 10 N.cm.
  Interventions: Other: Changing the implant surface; Radiation: Low Laser Radiation off; Procedure: Implant placement immediately after tooth extraction; Procedure: Installing the dental crown with early loading

INTERVENTIONS:
Radiation: Low Laser Radiation — One group will receive laser application to check if there is acceleration of healing.
  Arms: Implants GM Acqua surface, with LLLT.; Implants GM NeoPoros surface, with LLLT.
Other: Changing the implant surface — Changing the treatment surface of the dental implant to see if osseointegration occurs more quickly.
  Arms: Implants GM NeoPoros surface, with LLLT.; Implants NeoPoros surface, without LLLT.
Radiation: Low Laser Radiation off — This group will receive laser application off.
  Arms: Implants GM Acqua surface, without LLLT.; Implants NeoPoros surface, without LLLT.
Procedure: Implant placement immediately after tooth extraction — When the last alternative is tooth extraction, this will be done, and in the same surgical intervention the dental implant will be placed.
Procedure: Installing the dental crown with early loading — The installation of the dental crowns will be performed in a period of 6 to 8 weeks, after the dental implant has been installed.

SUMMARY:
Post-extraction implants are an alternative to traditional implant placement on completely healed bone, in order to reduce the number of surgical interventions, shorten treatment time, maintain bone architecture and thus provide better aesthetics. This study focuses on evaluating the results obtained by opting for different immediate placement of single dental implants protocols in a fresh alveolus, and its general objective is to compare implant stability and marginal bone loss (MBL) in implants installed post-extraction. For this, the investigators will placement Grand Morse Acqua or NeoPoros implants (Helix GM - Neodent, Curitiba, Brazil), in early loading protocols, with or without low level laser photobiomodulation (LLLT), in patients attending the Master of Oral Medicine, Oral Surgery and Implantology of the University of Santiago de Compostela for oral rehabilitation using osseointegrated single dental implants in the maxillary and/or mandibular region.

ELIGIBILITY:
Inclusion Criteria:

* Patients satisfying all inclusion criteria and none of the exclusion criteria will be informed verbally and in writing about the study and signed the informed consent form.
* The implant area is free of infection
* Patients without systemic pathology or medical and general contraindications that are absolute contraindications for surgical procedures;
* Adults who agree to take part in the study and signed the informed consent form.
* Smokers of less than 5 cigarettes/day.
* Not to be completely edentulous.
* Need for extraction of at least one tooth.
* Post-extraction bone area (fresh alveolus).
* Patients with sufficient bone height to obtain primary stability for implant installation (2 mm longer than the largest root).
* Edentulous areas with sufficient mesial-distal, buccolingual and interocclusal space for the placement of an anatomical restoration with a prosthetic space of at least 5 mm.

Exclusion Criteria:

* Immunosuppressed.
* Smokers of more than 5 cigarettes/day.
* Bleeding rate greater than 30 %.
* Presence of active or uncontrolled periodontal disease;
* Patients with less than 2 mm of keratinised gingiva.
* Implants with primary stability with ISQ < 50
* When this is not possible, assume a security margin to the inferior dental nerve of at least 1 mm.
* Previus history of local radiotherapy in the head and neck region.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Implant survival rate | 3 months
  After comparative of; Acqua/NeoPoros surface and LLLT/No LLLT application. Final total number.
Implant stability | 3 months
  Basal and 3 months postimplantation measured by Implant Stability Quotient (ISQ).
Marginal bone loss | 3 months
  Measured (mm) from the implant platform to the most coronal part of the peri-implant bone crest.

SECONDARY OUTCOMES:
Implant failure | 3 months
  To be assessed 3 months after surgery. Implant failure will be defined as implant failure when it is necessary to remove the implant due to implant mobility as a consequence of loss of osseointegration. Final total number.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Santiago de Compostela, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: Undecided
We will anonymize and categorize the clinical data of the patients to share the information with the other researchers of the group.